CLINICAL TRIAL: NCT07203729
Title: Trastuzumab Rezetecan (SHR-A1811) Versus Chemotherapy of Physician's Choice in Patients With HER2-Low Unresectable/Metastatic Breast Cancer Complicated With Visceral Crisis：A Randomized, Prospective, Open-Label Phase II Trial.
Brief Title: The Efficacy and Safety of Trastuzumab Rezetecan (SHR-A1811) in HER2-Low Unresectable/Metastatic Breast Cancer Patients With Visceral Crisis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ma Fei，MD, Chief Physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-117
Record Dates: First submitted 2025-09-25; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: HER2-Low Unresectable/Metastatic Breast Cancer Complicated With Visceral Crisis
Keywords: HER2-Low unresectable/metastatic breast cancer; Visceral Crisis; Antibody drug conjugates; Trastuzumab Rezetecan
MeSH Terms: conditions — Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; eribulin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1：Trastuzumab Rezetecan (Experimental)
  Interventions: Drug: Trastuzumab Rezetecan
- Arm 2：Chemotherapy of Physician's Choice (Active Comparator)
  Interventions: Drug: Chemotherapy of Physician's Choice

INTERVENTIONS:
Drug: Trastuzumab Rezetecan — Trastuzumab Rezetecan 4.8mg/kg, IV, Day 1, Q3W
  Arms: Arm 1：Trastuzumab Rezetecan
Drug: Chemotherapy of Physician's Choice — Chemotherapy of Physician's Choice, including nab-paclitaxel, Eribulin, Capecitabine
  Other Names: nab-paclitaxel; Eribulin; Capecitabine
  Arms: Arm 2：Chemotherapy of Physician's Choice

SUMMARY:
The goal of this clinical trial is to learn if Trastuzumab Rezetecan (SHR-A1811) is safe and tolerable for patients with HER2-Low unresectable/metastatic breast cancer complicated with visceral crisis. Participants will take Trastuzumab Rezetecan every three weeks, until disease progression or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years old and ≤75 years old;
* Pathologically confirmed HER2-Low unresectable or metastatic breast cancer;
* Investigators assess that the patient is at risk of rapid disease progression and presents signs, clinical symptoms, or laboratory abnormalities of visceral metastasis, including：a）Hepatic crisis: Rapid elevation of bilirubin > 1.5 × upper limit of normal (ULN) in the absence of Gilbert syndrome or biliary obstruction；b）Pulmonary crisis: Rapid exacerbation of dyspnea at rest, which is not relieved by pleural effusion drainage；c）Other visceral crises: Symptomatic visceral metastasis.
* Patients whom investigators deem to have indications for single-agent chemotherapy.
* Sufficient bone marrow function, defined as follows：a) Neutrophil count (ANC) ≥ 1,500/mm³ (1.5 × 10⁹/L)；b) Platelet count (PLT) ≥ 100,000/mm³ (100 × 10⁹/L)；c) Hemoglobin (Hb) ≥ 80 g/L；
* Patients who have received ≤ 1 line of chemotherapy in the advanced stage are permitted.
* Patients who have received endocrine therapy in the advanced stage are permitted.
* Previous treatment with CDK4/6 inhibitors is permitted.
* Previous or concurrent local treatment for symptom relief is permitted.
* For female subjects who are premenopausal or not surgically sterilized:

A serum pregnancy test must be performed within 7 days before the first dose of study drug, with a negative result. They must agree to either abstain from sexual activity or use a medically approved highly effective contraceptive method from the time of signing the informed consent form, throughout the study period, and for 1 year after the last dose of study drug.

* Patients must voluntarily participate in this study, sign the informed consent form, have good compliance, and be willing to cooperate with follow-up.

Exclusion Criteria:

* Have received treatment with new antibody-drug conjugates (ADCs) at any stage of breast cancer.
* Are deemed by the investigator as unsuitable for systemic chemotherapy.
* Have had other malignant tumors within the past 5 years, excluding cured carcinoma in situ of the cervix, cutaneous basal cell carcinoma, or cutaneous squamous cell carcinoma (patients with other malignant tumors that occurred more than 5 years before randomization and were cured solely by surgery are eligible for enrollment).
* Have undergone major surgical procedures or suffered significant trauma within 4 weeks prior to randomization, or are expected to undergo major surgical treatment.
* Have severe heart disease or cardiac discomfort, including but not limited to the following conditions：a) A history of heart failure or systolic dysfunction (left ventricular ejection fraction [LVEF] < 50%)；b) High-risk angina pectoris requiring treatment or cardiac arrhythmias；c) Clinically significant valvular heart disease；d) ECG findings indicating transmural myocardial infarction；e) Poorly controlled hypertension.
* Have a known history of allergy to any component of the drugs in this protocol.
* Have a history of immunodeficiency, including HIV infection, or other acquired or congenital immunodeficiency diseases.
* Have a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Have a known history of psychotropic substance abuse or drug addiction.
* Are pregnant or lactating women, or women of childbearing age who are unwilling to use effective contraceptive measures throughout the trial period and within 7 months after the last administration of the study drug.
* Have severe diseases, other comorbidities that would interfere with the planned treatment, or any other conditions that make them unsuitable for participation in this study (e.g., active hepatitis B, pulmonary infection requiring treatment).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2030-06-15 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From the start of treatment to 36 month
  Progression-Free Survival is defined as the time from randomization to first documented disease progression (PD) using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) or death from any cause, whichever occurred first. The PFS will be will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median PFS, hazard ratio with appropriate confidence intervals will be reported.

SECONDARY OUTCOMES:
Clinical Benefit Response (CBR) | From the start of treatment to 36 month
  CBR is percentage of participants with best (confirmed) PR or CR or SD for at least 6 months. PR or CR or SD is according to RECIST version 1.1. The CBR will be reported by percentage with each arms and appropriate confidence intervals.
Objective Overall Response Rate (ORR) | From the start of treatment to 36 month
  ORR is defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR. ORR was assessed by the investigator according to RECIST version 1.1 and is based on BOR, which is defined as best response recorded from start of study treatment until disease progression/recurrence or death. The ORR will be reported by percentage with each arms and appropriate confidence intervals.
Overall Survival (OS) | From the start of treatment to 36 month
  Overall Survival , defined as the time from the start of treatment to the date of death, regardless of the cause of death. The OS will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median OS, hazard ratio with appropriate confidence intervals will be reported.
Adverse events (AEs) | From the start of treatment to 36 month
  AEs were graded according to the National Cancer Institute's Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0. The type, grade and frequency of AEs will be reported.

IPD SHARING:
Plan to Share IPD: Undecided